CLINICAL TRIAL: NCT06451107
Title: Effectiveness of Specific Strength Training Combined With Static Stretching of the Posterior Neck in Office Workers With Chronic Neck Pain: A Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, María Santos, physiotherapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSP-2024
Record Dates: First submitted 2024-06-03; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain; Work Injury
Keywords: randomized controlled trial; Neck pain; exercise; Occupational Health
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The design will consist of a single-blind, randomized controlled trial, corresponding to an experimental longitudinal analytical study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strength training and static stretching (Experimental): The intervention will consist of a strength training program for the neck and shoulder muscles combined with static stretching of the neck.
  Interventions: Other: specific strength training with static neck stretching
- strength training (Active Comparator): The comparison group will only perform strength training.
  Interventions: Other: Specific Strength Training

INTERVENTIONS:
Other: specific strength training with static neck stretching — The intervention will consist of specific strength training composed of 5 exercises performed with dumbbells: front raises, lateral raises, reverse flies, shoulder shrugs, and wrist extensions. In addition to the following static stretches: stretching towards lateral flexion of the upper part of the trapezius muscle, the scalene muscles, and the sternocleidomastoid muscle on both sides; extension of the extensor muscles; flexion of the flexor muscles; and contralateral flexion and rotation combined with scapular depression of the scalene muscles and elevation of the scapula on both sides, holding each stretch for 10 seconds. This sequence of stretches will constitute one set, with 6 sets performed with a 30-second rest between sets, lasting 8 minutes. Therefore, the intervention will have a total duration of 28 minutes per session, conducting 3 sessions per week.
  Arms: strength training and static stretching
Other: Specific Strength Training — The intervention will consist of specific strength training comprised of 5 exercises using dumbbells: front raises, lateral raises, reverse flies, shoulder shrugs, and wrist extensions. Four sets will be performed, with a 1-minute rest between sets. Each exercise will be executed for 30 seconds, followed by a 25-second rest between exercises. Three 20-minute sessions will be conducted per week.
  Arms: strength training

SUMMARY:
Objective: To determine the effectiveness of strength training combined with stretching compared to specific strength training in office workers with chronic neck pain.

Methods: A single blind randomized clinical trial will be conducted. Participants will be adult of both sexes with sedentary office work and chronic neck pain.

The intervention will consist of a strength training program for the neck and shoulder muscles combined with static stretching of the neck, while the comparison group will only perform strength training. In addition, both groups will receive ergonomics guidelines.

Short-term, medium-term, and long-term evaluations will be performed using the Northwick Park Neck Pain Questionnaire (NPQ), Neck Disability Index (NDI), and Tampa Scale of Kinesiophobia (TSK).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 70 years.
* Workers from companies in the Community of Madrid.
* Sedentary employees who work at least 20 hours in the office.
* Subjects with nonspecific chronic neck pain.
* All individuals who have decided to participate voluntarily after having read and signed the patient information sheet and the informed consent form.

Exclusion Criteria:

* Arterial hypertension (systolic BP >160, diastolic BP >100) or cardiovascular diseases.
* Diagnosed metabolic disorders.
* Symptomatic disc herniation or severe cervical spine disorders.
* Postoperative conditions.
* History of severe trauma to the neck and shoulder region.
* Pregnancy.
* Subjects with a body mass index (BMI) greater than 29.9 kilograms per square meter (kg/m2).
* Presence of physical or mental impairments that prevent the correct execution of the interventions and/or their corresponding evaluation.
* Having undergone surgery in the previous six months.
* Participating in parallel research studies.
* Not having a permanent job position.
* Using two monitors.
* Using a laptop.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | It will be measured 4 times: before the start of the intervention, short-term (4 weeks), medium-term (2 months), and long-term (1 year).
  We will use the "Northwick Park Neck Pain Questionnaire", which consists of 9 questions with 5 statements of increasing difficulty. The minimum and maximum values are from 0 to 50 points. Higher scores indicate greater severity of neck pain.
Kinesiophobia | It will be measured 4 times: before the start of the intervention, short-term (4 weeks), medium-term (2 months), and long-term (1 year).
  We will use the "Tampa Scale for Kinesiophobia," which consists of 11 questions with 4 numeric options, ranging from 1 (completely disagree) to 4 (completely agree). The minimum and maximum values range from 17 to 68 points; higher scores indicate higher levels of kinesiophobia.
Neck Disability | It will be measured 4 times: before the start of the intervention, short-term (4 weeks), medium-term (2 months), and long-term (1 year).
  We will use the "Neck Disability Index," which consists of 10 questions with 6 statements of increasing difficulty. The values range from 0 to 50, where 0 indicates no disability and 50 indicates total disability.

CONTACTS AND LOCATIONS:
Overall Officials: María Santos, Principal Investigator — University of Alcala

IPD SHARING:
Plan to Share IPD: No